CLINICAL TRIAL: NCT04175847
Title: To Evaluate the Safety of RC88 for Injection in Patients With Advanced Malignant Solid Tumors,Multicenter, Open, Multi-cohort Extension of Efficacy and Pharmacokinetic Characteristics Phase I /IIa Clinical Study
Brief Title: A Phase I /IIa Study of RC88-ADC in Subjects With Advanced Malignant Solid Tumors
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: RemeGen Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RC88-C001
Record Dates: First submitted 2019-11-22; First posted 2019-11-25 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2025-12

CONDITIONS: Solid Tumor
MeSH Terms: interventions — Injections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- RC88 (Experimental)
  Interventions: Drug: RC88

INTERVENTIONS:
Drug: RC88 — Phase I:Participants will be allocated to one of the following dose groups: 0.1, 0.5, 1.0, 1.5, 2.0 and 2.5 mg/kg, and receive a treatment of RC88-ADC followed by 21 days of dose limited toxicity (DLT) observation period.
  Phase IIa indication exploration
  Other Names: RC88 for Injection

SUMMARY:
This was a multicenter, open, multi-cohort extended PHASE I/IIa study, consisting of 2 phases:Phase I (Phase I dose escalation) and Phase II (Phase IIa multi-cohort extension). The objective of this study was to evaluate safety, tolerability, pharmacokinetic characteristics, and initial efficacy in malignant pleural mesothelioma and MSLN in advanced malignant solid tumors.

DETAILED DESCRIPTION:
Phase I dose escalation phase：This study predicted a total of 6 dose groups, 0.1, 0.5, 1.0, 1.5, 2.0 and 2.5 mg/kg.

Phase IIa efficacy exploration phase:This phase is the multi-cohort indication expansion phase. Based on the data obtained in phase I, chose an appropriate dose continue to explore multi-cohort indications, including confirmed malignancy Pleural mesothelioma and MSLN expression were determined.

ELIGIBILITY:
Inclusion Criteria:

* Voluntary agreement to provide written informed consent.
* Age requirements ：phase I 18-70 (including 18 and 70) ,IIa ≥18 years old.
* Predicted survival ≥ 12 weeks.
* Phase I must be histologically or cytologically confirmed and have failed standard therapy (disease progression after treatment) or are intolerant, unable to receive, or nonexistent to standard care,Patients with partial advanced or metastatic malignant solid tumors;
* Phase II： Cohort 1：Advanced malignant mesothelioma； Cohort2：advanced ovarian carcinoma ；Cohort2 Other cancers that may benefit include pancreatic cancer, gastric adenocarcinoma, triple negative breast cancer, and lung adenocarcinoma
* Patients with malignant pleural mesothelioma were assessed using mRECIST criteria, and those with other cancers were assessed using RECIST V1.1 criteria.
* Mesothelin (MSLN) positive as confirmed by the central laboratory. Subject is able to provide specimens from primary or metastatic lesions for MSLN tests.
* Eastern Cooperative Oncology Group (ECOG) performance status score of 0 or 1.
* Adequate organ function, evidenced by the following laboratory results within 7 days prior to the study treatment:
* Cardiac ejection fraction ≥ 50 %. Hemoglobin ≥ 9g/dL; Absolute neutrophil count ≥ 1.5×10^9 /L Platelets ≥ 100×10^9 /L; Total bilirubin ≤ 1.5× ULN; AST and ALT ≤ 2.5×ULN and ≤ 5 x ULN with hepatic metastasis; Serum creatinine ≤1.5×ULN.
* All female subjects will be considered to be of child-bearing potential unless they are postmenopausal, or have been sterilized surgically.Female subjects of child-bearing potential must agree to use two forms of highly effective contraception. Male subjects and their female partner who are of child-bearing potential must agree to use two forms of highly effective contraception.
* Willing to adhere to the study visit schedule and the prohibitions and restrictions specified in this protocol.

Exclusion Criteria:

* Use of investigational drug or device within 4 weeks prior to study dosing
* Known hypersensitivity to the components of RC88-ADC.
* Toxicity of previous anti-tumor treatment not recovered to CTCAE Grade 0-1 (with exception of Grade 2 alopecia).
* Pericardial effusion or cardiac tamponade, or pleural or abdominal effusion with clinical symptoms that requires ongoing treatment.
* Has a history or current history of explosive, acute, chronic, recurrent or persistent myocarditis or pericarditis caused by any cause (eg, virus, tuberculosis, autoimmune disease, etc.)
* Ophthalmic screening is required: has a history of ocular lesions such as the cornea, limbus, conjunctiva, or eyelids (including but not limited to: corneal inflammation, corneal dystrophy, dry eye, meibomian gland dysfunction, uveitis, corneal endothelium Decompensation, glaucoma, iris corneal endothelial syndrome (ICE), etc.) can not be enrolled; has a ophthalmologists-confirmed current medical history of the cornea, limbus, conjunctiva, orbital lesions cannot be included;
* History of receiving any anti-cancer drug/biologic treatment within 4 weeks prior to trial treatment.
* History of major surgery within 4 weeks of planned start of trial treatment.
* Has received live virus vaccine within 4 weeks prior to study administration or planned to receive live virus vaccine during study .
* Currently known active infection with HIV or tuberculosis.
* Diagnosed with HBsAg , HBcAb positive and HBV DNA copy positive, or HCVAb positive.
* Has Unstable angina, coronary angioplasty, stent implantation,Coronary artery bypass grafting, serious arrhythmias requiring treatment (e.g., persistent ventricular tachycardia, ventricular fibrillation,Torsional ventricular tachycardia), QTc > 470 ms and long QT syndrome
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
* History of other malignancy within the previous 5 years, except for appropriately treated carcinoma in situ of the cervix, non-melanoma skin carcinoma, or cancers with a similar curative outcome as those mentioned above.
* known central nervous system metastases.
* Uncontrolled hypertension, diabetes, Interstitial lung Disease, or COPD;
* Pregnancy or lactation.
* Assessed by the investigator to be unable or unwilling to comply with the requirements of the protocol.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 198 (Actual)
Dates: Start 2020-04-14 (Actual); Primary Completion 2025-12-31 (Actual); Study Completion 2025-12-31 (Actual)

PRIMARY OUTCOMES:
Phase 1 Adverse events | From the day of ICF sign to 28 days after the day of the last treatment
  Adverse events was assessed by investigator(s) according to NCI-CTCAE v4.03
Phase 1 Maximum Tolerated dose of RC88 | 21 days after first treatment.
  The dose level in which >= 2 out of 6 patients have dose-limiting toxicity (DLT). The MTD is defined as the previous dose level.
Phase2 | 24 weeks
  ORR is evaluated by IRC

SECONDARY OUTCOMES:
Phase 1 Objective Response Rate (ORR) | 24 months
  Objective Response Rate was defined as the percentage of participants with a complete response (CR) or partial response (PR)
Phase 1 Progression Free Survival (PFS) | 24 months
  Progression-free Survival (PFS) (median) was determined using the number of months measured from the initial date of treatment to the date of documented progression, or the date of death (in the absence of progression) of participants. Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions.
Phase 1 and Phase2 Pharmacokinetics (PK) parameter for total antibody (TAb): Maximum concentration (Cmax) | Phase 1:Cycle 1 and Cycle 3 (each cycle is 21 days): pre-dose, 0.5 hour (hr), 1 hr, 1.5 hrs, 12 hrs, 24 hrs, 48 hrs, 72 hrs, 120 hrs, 168 hrs, 240 hrs (and 336 hrs) after start of infusion. Cycle 2: pre-dose.Phase2 （Whole test cycle）
  Cmax will be derived from the PK blood samples collected.
Phase 1 and Phase2 PK parameter for TAb: Time to maximum concentration (Tmax) | Cycle 1 and Cycle 3 (each cycle is 21 days): pre-dose, 0.5 hr, 1 hr, 1.5 hrs, 12 hrs, 24 hrs, 48 hrs, 72 hrs, 120 hrs, 168 hrs, 240 hrs (and 336 hrs) after start of infusion. Cycle 2: pre-dose.Phase2 （Whole test cycle）
  Tmax will be derived from the PK blood samples collected.
Phase 1 PK parameter for TAb: Area under the concentration-time curve (AUC) | Cycle 1 and Cycle 3 (each cycle is 21 days): pre-dose, 0.5 hr, 1 hr, 1.5 hrs, 12 hrs, 24 hrs, 48 hrs, 72 hrs, 120 hrs, 168 hrs, 240 hrs (and 336 hrs) after start of infusion. Cycle 2: pre-dose.
  AUC will be derived from the PK blood samples collected.
Phase 1 PK parameter for TAb: Trough concentration (Ctrough) | Cycle 1 and Cycle 3 (each cycle is 21 days): pre-dose, 0.5 hr, 1 hr, 1.5 hrs, 12 hrs, 24 hrs, 48 hrs, 72 hrs, 120 hrs, 168 hrs, 240 hrs (and 336 hrs) after start of infusion. Cycle 2: pre-dose.
  Ctrough will be derived from the PK blood samples collected.
Phase 1 PK parameter for TAb: Terminal or apparent terminal half-life (t1/2) | Cycle 1 and Cycle 3 (each cycle is 21 days): pre-dose, 0.5 hr, 1 hr, 1.5 hrs, 12 hrs, 24 hrs, 48 hrs, 72 hrs, 120 hrs, 168 hrs, 240 hrs (and 336 hrs) after start of infusion. Cycle 2: pre-dose.
  t1/2 will be derived from the PK blood samples collected.
Phase 1 PK parameter for TAb: Systemic clearance (CL) | Cycle 1 and Cycle 3 (each cycle is 21 days): pre-dose, 0.5 hr, 1 hr, 1.5 hrs, 12 hrs, 24 hrs, 48 hrs, 72 hrs, 120 hrs, 168 hrs, 240 hrs (and 336 hrs) after start of infusion. Cycle 2: pre-dose.
  CL will be derived from the PK blood samples collected.
Phase 1 PK parameter for antibody-drug conjugate (ADC): Cmax | Cycle 1 and Cycle 3 (each cycle is 21 days): pre-dose, 0.5 hr, 1 hr, 1.5 hrs, 12 hrs, 24 hrs, 48 hrs, 72 hrs, 120 hrs, 168 hrs, 240 hrs (and 336 hrs) after start of infusion. Cycle 2: pre-dose.
  Cmax will be derived from the PK blood samples collected.
Phase 1 PK parameter for ADC: Tmax | Cycle 1 and Cycle 3 (each cycle is 21 days): pre-dose, 0.5 hr, 1 hr, 1.5 hrs, 12 hrs, 24 hrs, 48 hrs, 72 hrs, 120 hrs, 168 hrs, 240 hrs (and 336 hrs) after start of infusion. Cycle 2: pre-dose.
  Tmax will be derived from the PK blood samples collected.
Phase 1 PK parameter for ADC: AUC | Cycle 1 and Cycle 3 (each cycle is 21 days): pre-dose, 0.5 hr, 1 hr, 1.5 hrs, 12 hrs, 24 hrs, 48 hrs, 72 hrs, 120 hrs, 168 hrs, 240 hrs (and 336 hrs) after start of infusion. Cycle 2: pre-dose.
  AUC will be derived from the PK blood samples collected.
Phase 1 PK parameter for ADC: Ctrough | Cycle 1 and Cycle 3 (each cycle is 21 days): pre-dose, 0.5 hr, 1 hr, 1.5 hrs, 12 hrs, 24 hrs, 48 hrs, 72 hrs, 120 hrs, 168 hrs, 240 hrs (and 336 hrs) after start of infusion. Cycle 2: pre-dose.
  Ctrough will be derived from the PK blood samples collected.
Phase 1 PK parameter for ADC: t1/2 | Cycle 1 and Cycle 3 (each cycle is 21 days): pre-dose, 0.5 hr, 1 hr, 1.5 hrs, 12 hrs, 24 hrs, 48 hrs, 72 hrs, 120 hrs, 168 hrs, 240 hrs (and 336 hrs) after start of infusion. Cycle 2: pre-dose.
  t1/2 will be derived from the PK blood samples collected.
PK parameter for ADC: CL | Cycle 1 and Cycle 3 (each cycle is 21 days): pre-dose, 0.5 hr, 1 hr, 1.5 hrs, 12 hrs, 24 hrs, 48 hrs, 72 hrs, 120 hrs, 168 hrs, 240 hrs (and 336 hrs) after start of infusion. Cycle 2: pre-dose.
  CL will be derived from the PK blood samples collected.
PK parameter for Monomethyl Auristatin E (MMAE): Cmax | Cycle 1 and Cycle 3 (each cycle is 21 days): pre-dose, 0.5 hr, 1 hr, 1.5 hrs, 12 hrs, 24 hrs, 48 hrs, 72 hrs, 120 hrs, 168 hrs, 240 hrs (and 336 hrs) after start of infusion. Cycle 2: pre-dose.
  Cmax will be derived from the PK blood samples collected.
PK parameter for MMAE: Tmax | Cycle 1 and Cycle 3 (each cycle is 21 days): pre-dose, 0.5 hr, 1 hr, 1.5 hrs, 12 hrs, 24 hrs, 48 hrs, 72 hrs, 120 hrs, 168 hrs, 240 hrs (and 336 hrs) after start of infusion. Cycle 2: pre-dose.
  Tmax will be derived from the PK blood samples collected.
PK parameter for MMAE: AUC | Cycle 1 and Cycle 3 (each cycle is 21 days): pre-dose, 0.5 hr, 1 hr, 1.5 hrs, 12 hrs, 24 hrs, 48 hrs, 72 hrs, 120 hrs, 168 hrs, 240 hrs (and 336 hrs) after start of infusion. Cycle 2: pre-dose.
  AUC will be derived from the PK blood samples collected.
PK parameter for MMAE: Ctrough | Cycle 1 and Cycle 3 (each cycle is 21 days): pre-dose, 0.5 hr, 1 hr, 1.5 hrs, 12 hrs, 24 hrs, 48 hrs, 72 hrs, 120 hrs, 168 hrs, 240 hrs (and 336 hrs) after start of infusion. Cycle 2: pre-dose.
  Ctrough will be derived from the PK blood samples collected.
PK parameter for MMAE: t1/2 | Cycle 1 and Cycle 3 (each cycle is 21 days): pre-dose, 0.5 hr, 1 hr, 1.5 hrs, 12 hrs, 24 hrs, 48 hrs, 72 hrs, 120 hrs, 168 hrs, 240 hrs (and 336 hrs) after start of infusion. Cycle 2: pre-dose.
  t1/2 will be derived from the PK blood samples collected.
PK parameter for MMAE: CL | Cycle 1 and Cycle 3 (each cycle is 21 days): pre-dose, 0.5 hr, 1 hr, 1.5 hrs, 12 hrs, 24 hrs, 48 hrs, 72 hrs, 120 hrs, 168 hrs, 240 hrs (and 336 hrs) after start of infusion. Cycle 2: pre-dose.
  CL will be derived from the PK blood samples collected.
Immunogenicity assessment | Cycle 1 to Cycle 3 (each cycle is 21 days): pre-dose, and 336 hrs after start of infusion (cycle 3 only).
  Assessment of anti-RC88 antibodies

CONTACTS AND LOCATIONS:
Locations (4):
- China (4):
  - National Cancer Center/Cancer Hospital, Chinese Academy of Medical Science and Peking Union Medical College, Beijing, Beijing Municipality
  - Henan Cancer Hospital, Zhengzhou, Henan
  - Drum Tower Hospital, Nanjing, Jiangsu
  - The First Hospital of Jilin University, Changchun, Jilin

IPD SHARING:
Plan to Share IPD: No